CLINICAL TRIAL: NCT05396638
Title: Characterization of Endocannabinoid and Endogenous Opioid Levels in Adolescents
Brief Title: Characterization of Endocannabinoid and Endogenous Opioid Levels in Adolescents With Cannabis Use Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Colorado Clinical & Translational Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20-0553
Record Dates: First submitted 2022-05-16; First posted 2022-05-31 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Cannabis Use

STUDY DESIGN:
Intervention Model Description: The contingency management (CM) procedure will consist of a four-week abstinence-based incentive program. At the initial visit, participants will be instructed to refrain from using cannabis for the next month and abstinence will be monitored by urine and saliva drug tests. Participants will be paid at each study visit for attendance and abstinence. CM payment rates for abstinence will revert to the initial payment level following a missed study visit or if THC levels rise or are detected by saliva drug screen, respectively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Contingency Management (Experimental): Abstinence will be rewarded following a contingency management (CM) payment scale.
  Interventions: Behavioral: Contingency Management

INTERVENTIONS:
Behavioral: Contingency Management — Participants will be paid for abstinence at each study visit.

SUMMARY:
This project seeks to learn more about the effects of cannabis use on the endocannabinoid system and endogenous opioid systems in adolescents to address a fundamental gap in knowledge and identify biomarkers that may help distinguish youth who relapse from youth who remain sober.

DETAILED DESCRIPTION:
Learning the effects of cannabis use on the endocannabinoid system and endogenous opioid systems in adolescents addresses a fundamental gap in knowledge and may identify biomarkers that help distinguish youth who relapse from youth who remain sober.

The specific aims of the project are to:

1. Measure endocannabinoid (eCB) and endogenous opioid (endorphin) levels in the blood of adolescents who use cannabis regularly and adolescents who never use cannabis. We expect eCB and endorphin levels to differ significantly in adolescents who use cannabis regularly compared to adolescents who do not.
2. Characterize circulating eCB and endorphin levels at baseline, during abstinence, and after natural resumption of cannabis use.
3. Collect data to evaluate cannabis craving and to test for association of craving with eCB and endorphin levels in adolescents who use cannabis regularly. We expect that larger changes in eCB and endorphin levels will be associated with higher craving scores.

ELIGIBILITY:
Inclusion Criteria:

1. 14 to 25 years of age.
2. Use cannabis at least twice a week for the past month.

Exclusion Criteria:

1. Refusal of valid written consent,
2. Current psychosis,
3. Obvious intoxication,
4. Current risk of suicide,
5. Violence sufficiently great to interfere with evaluation or to endanger evaluators,
6. Obvious intellectual deficiency as noted during the informed consent process, or inability of patient or family to comply with the study protocol.
7. Use of other illicit drugs in the past 90 days by self-report or detected by urine drug test.
8. Use of opioid medications for medical or recreational purposes currently or within the past 90 days.
9. Does not have access to an Internet connected devise or cannot use Zoom.

Ages: 14 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-13 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Cannabinoid levels in blood | Collected at Baseline
  Cannabinoid levels in blood: Our primary measure will be 11-nor-carboxy-Δ9-tetrahydrocannabinol (THCCOOH) concentrations in whole blood, which have been demonstrated to be a reliable quantitative measure of cannabis use over the past few weeks35. We will measure an additional 10 cannabinoids [THC, 11-hydroxy-THC, THC-glucuronide, cannabidiol (CBD), cannabinol (CBN), cannabigerol (CBG), cannabichromene (CBC), cannabidivarin (CBDV), tetrahydro-cannabivarin (THCV), and THCV-COOH]34, which will be visually inspected to identify potential secondary outcomes.
Cannabinoid levels in blood | Collected at Week 2
  Cannabinoid levels in blood: Our primary measure will be 11-nor-carboxy-Δ9-tetrahydrocannabinol (THCCOOH) concentrations in whole blood, which have been demonstrated to be a reliable quantitative measure of cannabis use over the past few weeks35. We will measure an additional 10 cannabinoids [THC, 11-hydroxy-THC, THC-glucuronide, cannabidiol (CBD), cannabinol (CBN), cannabigerol (CBG), cannabichromene (CBC), cannabidivarin (CBDV), tetrahydro-cannabivarin (THCV), and THCV-COOH]34, which will be visually inspected to identify potential secondary outcomes.
Cannabinoid levels in blood | Collected at Week 4
  Cannabinoid levels in blood: Our primary measure will be 11-nor-carboxy-Δ9-tetrahydrocannabinol (THCCOOH) concentrations in whole blood, which have been demonstrated to be a reliable quantitative measure of cannabis use over the past few weeks35. We will measure an additional 10 cannabinoids [THC, 11-hydroxy-THC, THC-glucuronide, cannabidiol (CBD), cannabinol (CBN), cannabigerol (CBG), cannabichromene (CBC), cannabidivarin (CBDV), tetrahydro-cannabivarin (THCV), and THCV-COOH]34, which will be visually inspected to identify potential secondary outcomes.
Cannabinoid levels in blood | Collected at Week 8
  Cannabinoid levels in blood: Our primary measure will be 11-nor-carboxy-Δ9-tetrahydrocannabinol (THCCOOH) concentrations in whole blood, which have been demonstrated to be a reliable quantitative measure of cannabis use over the past few weeks35. We will measure an additional 10 cannabinoids [THC, 11-hydroxy-THC, THC-glucuronide, cannabidiol (CBD), cannabinol (CBN), cannabigerol (CBG), cannabichromene (CBC), cannabidivarin (CBDV), tetrahydro-cannabivarin (THCV), and THCV-COOH]34, which will be visually inspected to identify potential secondary outcomes.
Endocannabinoid levels in blood | Collected at Baseline
  We will measure endocannabinoid (eCB) levels AEA and 2-AG, the primary eCBs, in whole blood.
Endocannabinoid levels in blood | Collected at Week 2
  We will measure endocannabinoid (eCB) levels AEA and 2-AG, the primary eCBs, in whole blood.
Endocannabinoid levels in blood | Collected at Week 4
  We will measure endocannabinoid (eCB) levels AEA and 2-AG, the primary eCBs, in whole blood.
Endocannabinoid levels in blood | Collected at Week 8
  We will measure endocannabinoid (eCB) levels AEA and 2-AG, the primary eCBs, in whole blood.

SECONDARY OUTCOMES:
Endorphin levels in blood | Collected at Baseline
  Endorphin levels in blood: Circulating beta Endorphin (b-EP) levels will be quantified using a commercially available enzyme-linked immunosorbent assay (ELISA) kit.
Endorphin levels in blood | Collected at Week 2
  Endorphin levels in blood: Circulating beta Endorphin (b-EP) levels will be quantified using a commercially available enzyme-linked immunosorbent assay (ELISA) kit.
Endorphin levels in blood | Collected at Week 4
  Endorphin levels in blood: Circulating beta Endorphin (b-EP) levels will be quantified using a commercially available enzyme-linked immunosorbent assay (ELISA) kit.
Endorphin levels in blood | Collected at Week 8
  Endorphin levels in blood: Circulating beta Endorphin (b-EP) levels will be quantified using a commercially available enzyme-linked immunosorbent assay (ELISA) kit.
Cannabis Craving | Collected at Baseline
  Cannabis craving: The Marijuana Craving Questionnaire (MCQ) will be used to assess cannabis craving.
Cannabis Craving | Collected at Week 2
  Cannabis craving: The Marijuana Craving Questionnaire (MCQ) will be used to assess cannabis craving.
Cannabis Craving | Collected at Week 4
  Cannabis craving: The Marijuana Craving Questionnaire (MCQ) will be used to assess cannabis craving.
Cannabis Craving | Collected at Week 8
  Cannabis craving: The Marijuana Craving Questionnaire (MCQ) will be used to assess cannabis craving.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No